CLINICAL TRIAL: NCT05957016
Title: Neoadjuvant Preoperative Arterial Intervention With Concurrent Chemoradiotherapy in Local Advanced Rectal Cancer
Brief Title: Neoadjuvant CIETAI With Concurrent Chemoradiotherapy in Local Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Dong Wang, dean of clinical oncology (fomer), Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIETAI-R
Record Dates: First submitted 2023-07-08; First posted 2023-07-24 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Rectal Cancer
Keywords: local advanced rectal cancer; PD-1 inhibitor; neoadjuvant
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- local advanced rectal cancer (Experimental): local advanced rectal cancer are defined as T3/4NanyM0 or T1-2N+M0
  Interventions: Procedure: CIETAI-R

INTERVENTIONS:
Procedure: CIETAI-R — 1. phase I: (1) Chemo-Immulo-embolization via Tumor Arterial, CIETAI: DSA guided tumor artery infusion of oxaliplatin 130 mg/m2+PD-1 inhibitor (Tirelizumab) 200mg, followed by gelatin sponge particles (350-560um) embolization
  2. phase II: Chemoradiotherapy: IMRT：45Gy/25f/5w+capecitabine 1000，po. Bid d1-14, q3w Tirelizumab)200mg ivggt, d1, q3w

SUMMARY:
To increase the efficacy of neoadjuvant PD-1/PD-1 checkpoint inhibitor in local advanced rectal cancer (LARC), we propose preoperative arterial infusion of Tirellizumab and oxaliplatin followed by tumor artery embolization with concurrent chemoradiotherapy as neoadjuvant regimen for LARC.

DETAILED DESCRIPTION:
Based our previous multi-center randomized controlled study (Preoperative arterial perfusion Chemo- embolization combined with radiotherapy for locally advanced rectal cancer, NCT03601156), the idea of "preoperative arterial chemo-immuno-embolization combined with radiotherapy for locally advanced rectal cancer (CIETAI-R)" was proposed. This is also the serial study of CIETAI that explore the efficacy of tumor arterial chemo-immuno-embolization in lung cancer, LARC, metastatic liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Local advanced Rectal cancer: stage T3/4NanyM0 or T1-2N+M0.
* Ages: 18 to 75.
* No previously received chemotherapy drugs and radiation therapy.
* ECOG score: 0 - 2.
* Appropriate organ function, as defined below:

(Hematology and blood biochemistry examination must be completed within 7 days before the registration date) i) White blood cell count ≥ 4,000/mm3. ii) Neutrophil count ≥ 1,500/mm3. iii) Hemoglobin ≥ 10 g/dL. iv) Platelet count ≥ 100,000/mm3. v) Total bilirubin ≤ 1.5 times the upper limit of normal (ULN). vi. Liver function Index (AST & ALT) ≤ 1.5 times the upper limit of normal (ULN).

vii. Serum creatinine ≤1.5 times the upper limit of normal or creatinine clearance ≥60 ml/min.

* Tolerance of orally administration of capecitabine.
* Can understand the study, have good compliance, cooperate with follow-up.

Exclusion Criteria:

* Severe allergic reaction to humanized antibodies or fusion proteins;
* Hypersensitivity to any component contained in contrast agent or granule embolic agent;
* Diagnosed with an immune deficiency or is receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 14 days prior to the first administration of the study, allowing the use of physiological doses of glucocorticoids (≤10mg/ day of prednisone or equivalent);
* Active, known, or suspected autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitaritis, vasculitis, nephritis, hypothyroidism, including, but not limited to, these diseases or syndromes). Subjects who have type 1 diabetes, hypothyroidism requiring hormone replacement therapy, skin conditions that do not require systemic treatment (e.g., vitiligo, psoriasis, or hair loss), or conditions that are not expected to recur in the absence of external triggers may be enrolled;
* Pre-existing severe heart disease, including congestive heart failure, uncontrolled high-risk arrhythmias, unstable angina pectoris, myocardial infarction, and severe heart valve disease;
* Active hepatitis B (HBV DNA ≥ 2000IU/ml or 104copies/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the lower limit of analysis).
* Active tuberculosis (TB) infection. Patients with a history of active tuberculosis infection within the previous 1 year should be excluded, even if they have been treated; Patients with a history of active tuberculosis infection more than 1 year ago should also be excluded unless the duration and type of antituberculosis therapy previously used is demonstrated to be appropriate.
* Brain metastases accompanied by symptoms or symptoms controlled for less than 2 months;
* Received major surgical treatment, open biopsy, or significant traumatic injury within 28 days prior to enrollment;
* Pregnant or lactating female patients (women of childbearing age must confirm that the pregnancy test is negative within 7 days before the first administration of the drug, if it is positive, ultrasound examination must be performed to rule out pregnancy), subjects of childbearing age refuse to accept contraceptive measures; Combined with other malignancies, except cured skin basal cell carcinoma or skin squamous cell carcinoma or in situ carcinoma of any other site
* Patients with any physical signs or history of bleeding, regardless of severity; Non-healing wounds, ulcers, or fractures were present in patients with any bleeding or bleeding events ≥CTCAE grade 3 during the 4 weeks prior to grouping;
* Arteriovenous thrombosis events within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism;
* Dementia, altered mental status or any mental illness that would prevent understanding or giving informed consent or completing the questionnaire
* Other serious concomitant diseases judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | 4 months

SECONDARY OUTCOMES:
disease-free survival (DFS) | 2 years
overall survival (OS) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang W, Qian C, Luo J, Chen C, Feng Y, Dai N, Li X, Xiao H, Yang Y, Li M, Li C, Wang D. First in human intraarterial delivery of tislelizumab for the treatment of pMMR locally advanced rectal cancer: A single-arm, open label, phase II clinical trial. Transl Oncol. 2024 Dec;50:102154. doi: 10.1016/j.tranon.2024.102154. Epub 2024 Oct 13. PMID 39405605